CLINICAL TRIAL: NCT00221533
Title: Relation Between Renin-Angiotensin Gene Polymorphisms, Plasma Adiponectin and Arterial Stiffness in Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Other Study IDs: 2005/196
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Vascular Diseases; Arterial Stiffness
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Relation between Renin-Angiotensin Gene Polymorphisms, Plasma Adiponectin and Arterial Stiffness in Renal Transplant Recipients

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years, extremes included
* Kidney transplants with or without other transplant organs
* Informed consent
* Stable clinical condition on the basis of a pre-trial physical examination, medical history, and the results of blood biochemistry and haematology tests

Exclusion Criteria:

* Pregnant, lactating females
* Recent (< 4 weeks) change in antihypertensive drug medication
* Current or recent (< 2 weeks) acute illness such as infection or bleeding
* Current treatment for malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-03; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Verbeke, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be